CLINICAL TRIAL: NCT04192487
Title: A Phase 4 Open Label Study to Assess the Safety and Effects of Crofelemer on the Gut Microbiome in Healthy Volunteers and in People Living With HIV/AIDS (PLWHA) With Non-Infectious Diarrhea
Brief Title: Effects of Crofelemer on the Gut Microbiome in Healthy Volunteers and in HIV+ Patients With Non-Infectious Diarrhea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Napo Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP 303-103
Record Dates: First submitted 2019-11-04; First posted 2019-12-10 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2020-11

CONDITIONS: Acquired Immunodeficiency Syndrome; Healthy Volunteers; HIV/AIDS; HIV Diarrhea; Human Immunodeficiency Virus
Keywords: Combination Antiretroviral Therapy (CART); CD4 Cell Count; Gut Microbiome; Non-Infectious Diarrhea; Diarrhea
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Healthy Volunteers (HIV-negative) (Experimental): Drug: crofelemer delayed-release tablets, 125 mg BID x 30 days
  Interventions: Drug: Crofelemer delayed-release tablets 125mg
- HIV+ Patients (Fully Suppressed, Viral Load < 50c/mL) (Experimental): Drug: crofelemer delayed-release tablets, 125mg BID x 30 Days
  Interventions: Drug: Crofelemer delayed-release tablets 125mg
- HIV+ Patients (Not fully suppressed viral load > 1000c/mL (Experimental): Drug: crofelemer delayed-release tablets, 125mg BID x 30 Days
  Interventions: Drug: Crofelemer delayed-release tablets 125mg

INTERVENTIONS:
Drug: Crofelemer delayed-release tablets 125mg — 1 crofelemer delayed-release tablet twice daily at least 8 hours apart for 30 days with or without meals.
  Other Names: Mytesi delayed-release tablets 125mg

SUMMARY:
This study is intended to evaluate:

1. Any changes in the gut microbiome from baseline compared to end of study in both healthy (HIV-negative) subjects and HIV+ patients with or without chronic diarrhea, following one month of treatment with crofelemer (Mytesi), delayed release 125 mg tablets twice daily (BID) following one month of treatment.
2. The safety and tolerability of crofelemer, (Mytesi) delayed release 125 mg tablets BID in healthy (HIV-negative) volunteers and HIV+ patients following one month of treatment.

DETAILED DESCRIPTION:
Mytesi ®(crofelemer) is an FDA-approved anti-diarrheal drug indicated for the symptomatic relief of non-infectious diarrhea in adult patients with HIV/AIDS on combination anti-retroviral therapy (CART). Crofelemer, a first-in-class intraluminally active, use-dependent chloride (Cl-) ion channel modulator that produces an antidiarrheal effect by reducing Cl- secretion and the accompanying high-volume fluid secretion into the GI lumen.

This Phase 4 trial will explore the induced gut microbiome changes in comparison to a group of normal healthy volunteers also receiving crofelemer delayed release 125 mg tablets twice daily for 30 days.

This is a non-randomized study. The study will enroll approximately 24 male or female subjects aged at least 18 years in three cohorts of approximately 8 subjects each.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary informed consent from the subject to be obtained in accordance with requirements of the Institutional Review Board (IRB) before any study-related activities are performed.
2. Body Mass Index (BMI) between 18 and 32 kg/m2 (both inclusive).
3. Females of child-bearing potential must have a negative serum pregnancy test result at Screening and a negative urine pregnancy test at Visit 2.

   Inclusion Criteria for Healthy, HIV-negative Volunteers
4. No history or evidence of clinically relevant medical disorders as determined by the investigator.
5. No history of chronic diarrhea or loose stools and/or non-specific incidence of acute diarrhea or loose stools between the Screening Visit and Baseline Visit 2 (Day 1).

   Inclusion Criteria applicable to all PLWHA subjects
6. Male and female patients receiving a stable CART for ≥ 4 weeks for HIV treatment.
7. Have a history of diarrhea (persistently loose stools despite periodic or regular use of antimotility medications) or ≥1 watery bowel movement per day (without periodic or regular use of antimotility drugs); i.e. - diarrhea for a continuous period of ≥1 month.

   Inclusion Criteria for PLWHA males and females receiving CART WITHOUT fully suppressed HIV RNA counts
8. CD4 counts >200/µL at the Screening Visit.
9. Plasma levels of HIV RNA greater than 1,000 copies/mL at the Screening Visit.

   Inclusion Criteria for PLWHA males and females receiving CART WITH fully suppressed HIV RNA counts
10. CD4 counts >400/µL inclusive at the Screening Visit.
11. Plasma levels of HIV RNA < 50 copies/mL at the Screening Visit.

Exclusion Criteria:

Applicable to ALL subjects

1. Any serious systemic disease or infection (other than HIV in PLWHA) that occurred within four weeks prior to Screening, as determined by the Investigator.
2. Patients with active bacterial or parasitic infections requiring antibiotics or antiparasitic agents will be excluded. Antibiotic or antiparasitic agents used for prophylaxis are acceptable until 7 days prior to treatment initiation.
3. Stool cultures that are positive for any pathogenic infection at screening visit.
4. Clinically significant cardiovascular disease will include:

   1. History of stroke, transient ischemic attack, or myocardial infarction within 6 months prior to Screening.
   2. History of or currently have New York Heart Association Class III-IV heart failure prior to Screening.
5. Female subject who is pregnant or breast-feeding or intends to become pregnant or is of childbearing potential and not using adequate contraceptive methods.
6. Subject has participated in another clinical study, involving an Investigational Product or an Investigational Device use in the past 1 month prior to commencement of this study.
7. Use of Mytesi (crofelemer) within 4 weeks of the Screening Visit Applicable to ALL HIV-negative subjects
8. Positive for Human Immunodeficiency Virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), hepatitis B core antibody or hepatitis C antibodies (HepCAb).
9. Presence or history of cancer within the past five years except for adequately treated localized basal cell skin cancer or in situ uterine cervical cancer.
10. Chronic diarrhea or loose stools requiring antimotility medications including, but not limited to loperamide, diphenoxylate/atropine, tincture opium and/or octreotide within 2 weeks of the Screening Visit.

    Applicable to ALL PLWHA subjects
11. HIV Patients with infectious diarrhea identified by either stool culture

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 17 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Changes in gut microbiome | Screening (Visit 1/Day -21) to end of Study Visit 4 (Day 60)
  Stool microbiomes will be evaluated to compare the differences in the stool microbiome at Visits 2, (Day 1) Visit 3 (Day 30) and Visit 4 (Day 60) using a proprietary microbiome statistical tool (μScope) and R statistical computing and graphics software.

SECONDARY OUTCOMES:
Evaluation of reduction in the number of watery BMs | From baseline (Day -7) to end of study (Day 60)
  Defined as a score of 6 or 7 on the Bristol Stool Scale
Assessment of changes in Daily GI symptom Scale (DGIS) | From baseline (Day -7) to end of study (Day 60)
  Daily presence or absence of abdominal pain, bloating, gurgling, flatulence, and bowel incontinence

CONTACTS AND LOCATIONS:
Overall Officials: David Smith, MD, Principal Investigator — Integrium Clinical Research
Locations (3):
- United States (3):
  - Orange County Research Center, Tustin, California
  - Healthcare Advocates International, Stratford, Connecticut
  - The Research Institute, Springfield, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siddiqui U, Bini EJ, Chandarana K, Leong J, Ramsetty S, Schiliro D, Poles M. Prevalence and impact of diarrhea on health-related quality of life in HIV-infected patients in the era of highly active antiretroviral therapy. J Clin Gastroenterol. 2007 May-Jun;41(5):484-90. doi: 10.1097/01.mcg.0000225694.46874.fc. PMID 17450031
- [Background] Cello JP, Day LW. Idiopathic AIDS enteropathy and treatment of gastrointestinal opportunistic pathogens. Gastroenterology. 2009 May;136(6):1952-65. doi: 10.1053/j.gastro.2008.12.073. Epub 2009 May 7. PMID 19457421
- [Background] MacArthur RD, DuPont HL. Etiology and pharmacologic management of noninfectious diarrhea in HIV-infected individuals in the highly active antiretroviral therapy era. Clin Infect Dis. 2012 Sep;55(6):860-7. doi: 10.1093/cid/cis544. Epub 2012 Jun 14. PMID 22700829
- [Background] Tradtrantip L, Namkung W, Verkman AS. Crofelemer, an antisecretory antidiarrheal proanthocyanidin oligomer extracted from Croton lechleri, targets two distinct intestinal chloride channels. Mol Pharmacol. 2010 Jan;77(1):69-78. doi: 10.1124/mol.109.061051. Epub 2009 Oct 6. PMID 19808995
- [Background] Macarthur RD, Hawkins TN, Brown SJ, Lamarca A, Clay PG, Barrett AC, Bortey E, Paterson C, Golden PL, Forbes WP. Efficacy and safety of crofelemer for noninfectious diarrhea in HIV-seropositive individuals (ADVENT trial): a randomized, double-blind, placebo-controlled, two-stage study. HIV Clin Trials. 2013 Nov-Dec;14(6):261-73. doi: 10.1310/hct1406-261. PMID 24334179